CLINICAL TRIAL: NCT05935891
Title: A Feasibility Study of Topical Cannabinoids for Treatment of Aromatase Inhibitor-Associated Musculoskeletal Syndrome (AIMSS) in Adults With Hormone Receptor-Positive Breast Cancer (CanAroma)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIMSS
Record Dates: First submitted 2023-06-15; First posted 2023-07-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Musculoskeletal Syndrome

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to CBD-dominant (Violet) and THC-dominant (Red XS) balms.
Who Masked: Outcomes Assessor
Masking Description: Patients will be informed as to which product they are using.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Violet (Experimental): Patients receiving CBD-dominant balm
  Interventions: Drug: CBD-dominant
- Red Xs (Experimental): Patients receiving THC-dominant balm
  Interventions: Drug: THC dominant

INTERVENTIONS:
Drug: CBD-dominant — product contains 2210 mg CBD and less than 0.3% THC per 1.5 ounce jar. Patients will be provided a 2-week supply of creams (3 jars for each 14 day interval) by Vireo Health, according to the randomization arm. Patient will be instructed to apply the topical products using the 1.25cc spoon provided (there are approximately 35 scoops per 1.5oz jar). The patient will apply one scoop of cream to the back of each hand and then rub into the entire hand, wrist, and all fingers. After the 14 day assessment, patients will be transitioned to a two-week open label extension that allows them to choose their preference of either Red XS or Violet cream at no cost.
  Arms: Violet
Drug: THC dominant — contains 375mg THC and less than 20mg CBD per 1.5 ounce jar. Patients will be provided a 2-week supply of creams (3 jars for each 14 day interval) by Vireo Health, according to the randomization arm. Patient will be instructed to apply the topical products using the 1.25cc spoon provided (there are approximately 35 scoops per 1.5oz jar). The patient will apply one scoop of cream to the back of each hand and then rub into the entire hand, wrist, and all fingers. After the 14 day assessment, patients will be transitioned to a two-week open label extension that allows them to choose their preference of either Red XS or Violet cream at no cost.
  Arms: Red Xs

SUMMARY:
Aromatase inhibitors (AIs) are commonly used for post-menopausal women with hormone-positive breast cancer. Compared to tamoxifen, AIs improve breast cancer recurrence rates and lower 10-year breast cancer mortality. Unfortunately, nearly 2 out of 3 women with estrogen-receptor positive breast cancer treated with AIs experiences AIMSS, such as arthralgia, joint stiffness, and bone pain, and 30% of women with AIMSS report severe pain. AIMSS leads to poor adherence with therapy and discontinuation of therapy in up to 20% of patients. Despite the large number of women affected, current therapeutic interventions have shown only limited efficacy in improving AIMSS. Therefore, the presence of AIMSS may negatively impact breast cancer recurrence and survival. In this current trial, the plan is to utilize topical cannabinoid creams from Vireo Health that have been tested for potency and purity. Two distinct products with different THC/CBD ratios will be provided to patients at no cost; a) a THC-dominant cream (Red XS Balm with 375mg/jar and <20mg of CBD) and b) a CBD-dominant cream (Violet Balm with 2210mg CBD/jar and <0.3% THC). The study will explore the feasibility of doing larger, placebo controlled trials by first ensuring adequate patient interest, acceptable tolerability/safety of cream utilization, and preliminary efficacy measures. All patients completing assessments through day 14 will be allowed to choose either Red XS or Violet creams for an additional 2-week extension period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above at the time of signing the informed consent form.
* Histologically proven diagnosis of stage I-III invasive breast cancer.
* Currently taking prescribed dose of an aromatase inhibitor (e.g., anastrazole, letrozole, exemestane) for at least 60 days with a plan to continue for at least 4 weeks after time of consent.
* Initiated AI therapy must have been within 48 months at time of consent.
* Experiencing AIMSS in hands and/or wrists for at least 4 weeks prior to time of consent.
* Patients must have reported a score of 4 or higher on at least one of the four M-SACRAH questions regarding pain and stiffness in hands and/or wrists over the past 7 days. Patients experiencing AIMSS symptoms in other joints are eligible, but must have pain in hands and/or wrists.
* Must be willing and able to comply with study visits and procedures.
* Must be willing to be registered in the Minnesota Medical Cannabis Program (MMCP).
* Must meet qualifications for the Minnesota Medical Cannabis

Program (MMCP). This includes:

1. Must have a qualifying condition, as per MMCP requirements, that is certified by a Health Care Practitioner.
2. Must be a Minnesota resident.

Exclusion Criteria:

* The patient is currently using or has used cannabinoids within 4 weeks of time of consent.
* Active skin lesions on hands/wrists that the investigator feels could impair absorption of cannabinoid cream or lead to increased toxicity (e.g., psoriasis, cellulitis, cutaneous lupus erythematosus, hand-foot syndrome).
* Plan to start or increase doses of other analgesics aimed at improving AIMSS symptoms (e.g., duloxetine, non-steroidal anti- inflammatories, acetaminophen, opioids). Of note, patients are eligible if they have remained on stable doses of AIMSS related medications for 4 weeks prior to time of consent and do not plan to escalate the dose.
* Current or planned initiation of acupuncture to arms, wrists or hands within study period.
* Any known or suspected hypersensitivity to topical cannabinoids.
* Any condition that the investigator believes would interfere with the ability to provide informed consent, comply with the study protocol, or would put the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
subject recruitment rate | 4 weeks
  percentage of participants actually recruited out of anticipated
subject retention rate | 4 weeks
  percentage of participants who completed the study

SECONDARY OUTCOMES:
change in Brief Pain Inventory Short Form (BPI-SF) scores | 2 weeks and 4 weeks
  worst pain, average pain, pain interference with general activity minimum value is zero equals no pain and maximum value is 10 equals pain as bad as you can imagine and the higher the score the worse the outcome.
tolerability of topical medical cannabis creams | 2 weeks and 4 weeks
  documenting patient adherence to dosing protocol through a Patient Topical Cannabis Dosing Diary.
  This is a document where the patient records the date, time, to which hands the dose was applied and if the dose was missed.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Blaes, MD,MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States